CLINICAL TRIAL: NCT00154167
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of NV-101 in Dental Patients
Brief Title: Safety and Efficacy Study of NV-101 in Dental Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novalar Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NOVA 03-001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Soft Tissue Anesthesia (Numbness)
MeSH Terms: conditions — Hypesthesia

INTERVENTIONS:
Drug: NV-101 (phentolamine mesylate solution)

SUMMARY:
The purpose of this study was:

* to determine if NV-101 accelerates recovery from numbness compared to placebo
* to evaluate safety of NV-101

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, multi-center study. One hundred twenty-two patients aged 10-58 requiring treatment with one of four routine dental procedures were enrolled. The investigators were licensed dentists in private practice. Each patient received one or more conventional injections of either articaine with epinephrine, lidocaine with epinephrine, prilocaine with epinephrine, or mepivacaine with levonordefrin. Local anesthetics were injected into no more than 2 sites. Injections of local anesthetic placed within 4mm of each other constituted the same site. The injection(s) of study drug were made at or near the completion of the dental procedure and were required to be not earlier than 20 minutes after, and not later than 70 minutes after, the most recent injection of local anesthetic. Patients received an injection of study drug (1.8 mL) in each site at which local anesthetic had been injected (i.e. no more than 2 sites).

Patients self-evaluated the return of normal sensation in the lip, tongue, nose, and chin by palpations at 5-minute intervals beginning 1 minute before the study drug injection and continuing for a minimum of 3 hours and until they achieved the return of normal sensation in lip, tongue, nose, and chin.

Safety was assessed by the use of a Holter monitor, vital signs, pain ratings, and physical examinations including oral cavity examinations.

ELIGIBILITY:
Inclusion Criteria:

* Between 10-65 years of age
* Body weight between 35 to 110 kg
* Healthy as determined by the Investigator based on medical history, physical examination, and 12 Lead ECG
* Clinical laboratory tests within the reference ranges or within clinically acceptable limits according to the Investigator
* Normal lip, nose, chin, and tongue sensations
* Women of childbearing potential must have agreed to use barrier contraception for the duration of the study (Women of childbearing potential included all women except for those who are premenstrual, whose menstrual periods have not occured for greater than or equal to one year after menopause, who are surgically sterilized, or who have had a hysterectomy)
* Can understand and sign the informed consent document, can communicate with the investigator, and can understand and comply with the requirements of the protocol

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, or connective tissue disease or disorder
* Clinically relevant surgical history
* History of alcoholism and/or drug abuse within the past 5 years
* Significant infection or known inflammatory process including viral infections
* Required prophylactic antibiotics for SBE (infectious endocarditis)
* Had acute gastrointestinal symptoms at screening and/or baseline
* Allergies to any of the following: lidocaine/epinephrine, articaine/epinephrine, prilocaine/epinephrine, bisulfites or metasulfites, or phentolamine
* Had used any investigational drug and/or participated in any clinical trial within 30 days of baseline
* Used pain relievers 24 hours prior to anesthetic administration
* Required the use of nitrous oxide or sedatives to perform the scheduled, eligible dental procedure
* Pregnancy, attempting to conceive,or lactating
* Used decongestants or other drugs with vasoactive moieties within 24 hours prior to anesthetic administration

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122
Dates: Start 2003-02; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Overall Officials: Royce Morrison, MD, Principal Investigator — Northwest Kinetics
Locations (1):
- Northwest Kinetics, Tacoma, Washington, United States